CLINICAL TRIAL: NCT01438723
Title: The Metformin in CABG (MetCAB) Trial
Brief Title: The Metformin in Coronary Artery Bypass Graft (CABG) (MetCAB) Trial
Acronym: MetCAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MetCAB; 2011-000099-33 (EudraCT Number)
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2011-11

CONDITIONS: Cardiovascular Disease; Ischemic Heart Disease
Keywords: ischemia reperfusion injury; CABG; metformin; Hs-troponin-I
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Ischemia; Reperfusion Injury | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin (Experimental)
  Interventions: Drug: Metformin
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — prior to CAGB surgery 3 day treatment with metformin 500 mg three times a day
  Other Names: Glucophage
  Arms: metformin
Drug: Placebo — prior to CABG surgery 3 day treatment with placebo capsules three times a day
  Arms: placebo

SUMMARY:
Rationale:

In patients with a myocardial infarction, occlusion of a coronary artery induces myocardial ischemia and cell death. If untreated, the area of myocardium exposed to this interruption in blood supply, will largely become necrotic. The only way to limit final infarct size, is timely reperfusion of the occluded artery. Paradoxically, however, reperfusion itself can also damage myocardial tissue and contribute to the final infarct size ("reperfusion injury"). Also during coronary artery bypass grafting (CABG), the myocardium is exposed to ischemia and reperfusion, which will induce cell death. Indeed, postoperatively, the plasma concentration of troponin I, a marker of cardiac necrosis, is increased, and associated with adverse outcome. The anti-hyperglycaemic drug metformin has been shown in preclinical studies to be able to reduce ischemia-reperfusion injury and to limit myocardial infarct size. Moreover, metformin therapy improves cardiovascular prognosis in patients with diabetes mellitus. Paradoxically, in patients with diabetes, current practice is to temporarily stop metformin before major surgery for the presumed risk of lactic acidosis, which is a rare complication of metformin. However, here is no evidence that this practice benefits the patient. The investigators hypothesize that pretreatment with metformin can reduce myocardial injury in patients undergoing elective CABG surgery

ELIGIBILITY:
Inclusion Criteria:

* Acceptation for CABG with or without concomitant valve surgery
* Informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Diabetes mellitus
* Renal dysfunction (MDRD < 60 ml/min)
* Elevated liver enzymes (ALAT > 3 times upper limit of reference range)
* Treatment with dipyridamole or xanthine derivatives
* Recent myocardial infarction (<2 weeks before inclusion)
* Off-pump surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Hs-Troponin-I | within 24 hours after CABG
  high sensitive cardiac troponin-I

SECONDARY OUTCOMES:
Post operative occurrence of arrhythmias | within 24 hours after CABG
Duration of inotropic support | within two days after CABG
Time to detubation | within two days after CABG
Post-ischemic recovery of contractile function of atrial trabeculae | until 4 hours after harvesting

CONTACTS AND LOCATIONS:
Locations (1):
- RUNMC, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] El Messaoudi S, Nederlof R, Zuurbier CJ, van Swieten HA, Pickkers P, Noyez L, Dieker HJ, Coenen MJ, Donders AR, Vos A, Rongen GA, Riksen NP. Effect of metformin pretreatment on myocardial injury during coronary artery bypass surgery in patients without diabetes (MetCAB): a double-blind, randomised controlled trial. Lancet Diabetes Endocrinol. 2015 Aug;3(8):615-23. doi: 10.1016/S2213-8587(15)00121-7. Epub 2015 Jul 12. PMID 26179504
- [Derived] Riksen NP, el Messaoudi S, Rongen GA. It takes more than one CAMERA to study cardiovascular protection by metformin. Lancet Diabetes Endocrinol. 2014 Feb;2(2):105-6. doi: 10.1016/S2213-8587(13)70207-9. Epub 2014 Feb 3. No abstract available. PMID 24622709